CLINICAL TRIAL: NCT00336505
Title: A Double-Blinded, Randomized, Parallel Group, Multi-Center, Multi-National Comparative Study of the Safety and Efficacy of Cethromycin 300 mg QD to Clarithromycin (BIAXIN® Filmtab®) 250 mg BID for the Treatment of Community-Acquired Pneumonia in Adults
Brief Title: Study Comparing the Safety and Efficacy of Cethromycin to Clarithromycin for the Treatment of Community-Acquired Pneumonia (CAP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Advanced Life Sciences, Inc. (Industry)
Responsible Party: David Eiznhamer, PhD, Executive Vice President, Clinical Development, Advanced Life Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL05-001
Record Dates: First submitted 2006-06-09; First posted 2006-06-13 (Estimated); Results first posted 2010-02-26 (Estimated); Last update posted 2010-02-26 (Estimated); Status verified 2010-01

CONDITIONS: Pneumonia
Keywords: Pneumonia; Respiratory; Infection; Infectious; Advanced; Life; Sciences; Lung; Pulmonary; Cethromycin; Restanza; Clarithromycin; Biaxin
MeSH Terms: conditions — Pneumonia; Infections; Communicable Diseases | interventions — cethromycin; Clarithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clarithromycin (Active Comparator)
  Interventions: Drug: Clarithromycin
- Cethromycin (Experimental)
  Interventions: Drug: Cethromycin

INTERVENTIONS:
Drug: Cethromycin — Cethromycin 300 mg once per day (QD) for 7 days, administered orally
  Other Names: Restanza; ABT-773
  Arms: Cethromycin
Drug: Clarithromycin — Clarithromycin 250 mg twice per day (BID) for 7 days, administered orally
  Other Names: Biaxin; Klacid; Klaracid
  Arms: Clarithromycin

SUMMARY:
The purpose of this study is to compare the efficacy of cethromycin to clarithromycin for the treatment of mild to moderate community-acquired pneumonia (CAP).

DETAILED DESCRIPTION:
Lower respiratory tract infections remain one of the leading causes of death worldwide. Increasing rates of antibiotic resistance and newer, more pervasive pneumonia-causative pathogens contribute to this statistic. Currently available macrolide antibiotics for the treatment of community-acquired pneumonia are slowly losing effectiveness, resulting in the need to develop newer drugs to fight resistant infections. In this study, we compare the safety and efficacy of a common macrolide, clarithromycin, to a new ketolide, cethromycin.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory male or female, 18 years of age or older
* If female, non-lactating and at no risk or pregnancy (post-menopausal or must use adequate birth control)
* Positive Chest X-ray consistent with diagnosis of bacterial pneumonia
* Must be a suitable candidate for oral antibiotic therapy and must be able to swallow capsules intact
* Recent history of respiratory illness consistent with the clinical signs and symptoms of bacterial CAP
* Must be able to produce sputum

Exclusion Criteria:

* Prior hospitalization within previous 4 weeks
* Residence at a chronic care facility
* Active tuberculosis (or other mycobacterial infection, empyema, lung abscess, pulmonary embolism, pulmonary edema, cystic fibrosis, tumor (primary or metastatic) involving the lung, bronchial obstruction, a history of post-obstructive pneumonia (chronic obstructive pulmonary disease [COPD] is not exclusionary), known or suspected Pneumocystis carinii pneumonia
* Treatment with long-acting antimicrobial agents within the last 4 weeks, treatment with ceftriaxone, azithromycin or dirithromycin antibiotic within the last 7 days, or subjects who have received more than 24 hours of treatment with other antibiotics within 7 days prior to study drug administration
* Any infection which requires the use of a concomitant antimicrobial agent
* History of hypersensitivity or allergic reactions to macrolide, ketolide, quinolone, azalide or streptogramin antimicrobials
* Treatment with another investigational drug within the last 4 weeks
* Females who are pregnant or lactating
* Subjects with known significant renal or hepatic impairment or disease
* Subjects with a history of impaired renal function
* Evidence of uncontrolled clinically significant cardiovascular, pulmonary, metabolic, gastrointestinal, neurological or endocrine disease, malignancy, or other abnormality (other than the disease being studied)
* Subjects who would require parenteral antimicrobial therapy for the treatment of pneumonia
* Any underlying disease or condition that would interfere with the completion of the study procedures and evaluations or absorption of the study drug
* Currently receiving or are likely to require any of the following medications during the period between 2 weeks prior to Evaluation 1 and within 24 hours after the last dose of study drug: astemizol (Hismanal®) or pimozide (Orap®)
* Currently receiving or are likely to require any of the following during the period from Evaluation 1 and within 24 hours after the last dose of study drug: theophylline or theophylline analogues (unless adequately monitored), carbamazepine, dexamethasone, phenobarbital, phenytoin, St. John's Wort, lamotrigine, troglitazone, warfarin and digitalis glycoside. Other barbiturates may be used with careful monitoring
* Subjects who are currently receiving or who are likely to require any of the following medications during the period between Evaluation 1 and 4: other systemic antibiotic therapy, rifampin or rifabutin
* Immunocompromised subjects, subjects receiving immunosuppressive agents, subjects with known human immunodeficiency virus (HIV) infections and history of acquired immune deficiency syndrome (AIDS) defining conditions or CD4+ T-lymphocyte count <200.
* Subject with known or suspected central nervous system (CNS) disorder that predisposes them to seizures/lower seizure threshold (e.g., severe cerebral arteriosclerosis, epilepsy)
* Previous treatment with cethromycin
* Subjects with signs of septic shock (e.g., mental confusion, severe hypoxemia, severe hypotension, any other condition requiring intensive care unit [ICU] admission)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 584 (Actual)
Dates: Start 2005-12; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A. Eiznhamer, PhD, Study Director — Advanced Life Sciences
Locations (3):
- United States (3):
  - CANADA - Advanced Life Sciences, Woodridge, Illinois
  - SOUTH AFRICA - Advanced Life Sciences, Woodridge, Illinois
  - USA - Advanced Life Sciences, Woodridge, Illinois

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited globally from January 2006 through October 2007.
Pre-assignment Details: In each treatment arm, one subject was enrolled and randomized to a blinded treatment but discontinued from study prior to administration of the first dose of drug. Thus, while official enrollment totalled 584 subjects, only 582 were randomized and dosed with blinded study drug.
Groups:
- Cethromycin: 300 mg once per day (QD) for 7 days, administered orally
- Clarithromycin: 250 mg twice per day (BID) for 7 days, administered orally
Period: Overall Study
Arm/Group | Cethromycin | Clarithromycin
Started | 291 (All subjects who were randomized and dosed.) | 291 (All subjects who were randomized and dosed.)
Completed | 254 (Number of subjects completing the test of cure (TOC) visit.) | 264 (Number of subjects completing the test of cure (TOC) visit.)
Not Completed | 37 | 27
Not completed — Adverse Event | 10 | 9
Not completed — Lack of Efficacy | 8 | 4
Not completed — Lost to Follow-up | 7 | 4
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Other | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cethromycin | Clarithromycin | Total
Number analyzed (Participants) | 291 | 291 | 582
Age Continuous [Mean (Standard Deviation); unit: years] — All subjects who were randomized and dosed.
  years | 48.6 (14.5) | 50.3 (16.3) | 49.5 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants] — All subjects who were randomized and dosed.
  Participants
    Female | 140 | 143 | 283
    Male | 151 | 148 | 299

OUTCOME MEASURES:

1. Primary Outcome: Clinical Cures in the Intent to Treat Population
Description: Investigators evaluated subjects for a clinical response of cure, failure, or indeterminate. Cure: Improvement or return to preinfection state or lack of progression of all pulmonary infiltrates, and resolution of all signs/symptoms present at enrollment. Failure: Persistence or worsening of signs/symptoms, the need for additional antibiotic, new pulmonary infection, progression of the chest radiograph, or death due to pneumonia. Indeterminate: Evaluation was not possible (lost to follow up, adverse event, major protocol violation). Indeterminates default to failure for analysis.
Time Frame: Test of Cure Visit, defined as 14-22 days after the first dose of study drug.
Population: The Intent to Treat Population is defined as all subjects with a confirmed diagnosis of community acquired pneumonia who took at least one dose of study medication. Subjects without a radiologist-confirmed chest X-ray for pneumonia were not included in the efficacy populations.
Measure: Number; unit: Participants
Arm/Group | Cethromycin | Clarithromycin
Number analyzed (Participants) | 261 | 254
Participants
  Clinical Cures | 217 | 206
  Clinical Failures | 14 | 13
  Indeterminates | 30 | 35
Statistical Analysis 1: Comparison: Cethromycin vs Clarithromycin; The rate of clinical cure in each treatment group was calculated (number of cures/number of patient eligible for analysis). Non-inferiority will be demonstrated when the lower limit of the two-sided 95% confidence interval for the difference in the clinical cure rate at the Test-of-Cure visit between treatment groups (Cethromycin -Clarithromycin) is greater than delta, and includes zero, for both Per-Protocol (PP) and Intent-to-Treat (ITT) analyses; Test type: Non-Inferiority or Equivalence — Delta will be determined by the highest clinical cure-rate between the Cethromycin treatment group and the Clarithromycin treatment group, as follows: Greater than or equal to 90%, delta = -10%; Greater than or equal to 80% and less than 90%, delta = -15%, Greater than or equal to 70% and less than 80%, -20%); p = 0.5667, Fisher Exact; Mean Difference (Net) = 2.0, 95% CI 2-sided [-4.8 to 8.9]

2. Secondary Outcome: Bacteriologic Cures in the Intent to Treat Population
Description: All bacteriologically evaluable subjects (ie., the subject had at least one, protocol-defined evaluable pathogen) who demonstrated eradication of all evaluable pathogens (S. pneumoniae, S. aureus, H. influenzae, M. catarrhalis, M. pneumoniae, C. pneumoniae, L. pneumophila).
Time Frame: Test of Cure Visit, defined as 14-22 days after the first dose of study drug.
Population: Includes all Intent to Treat subjects that were bacteriologically evaluable (ie., subjects with at least 1 evaluable pathogen) who showed eradication of all evaluable pathogens.
Measure: Number; unit: Participants
Arm/Group | Cethromycin | Clarithromycin
Number analyzed (Participants) | 81 | 85
Participants
  Bacteriologic Cures | 73 | 73

3. Primary Outcome: Clinical Cures in the Per Protocol Clinically Evaluable Population
Description: as for outcome 1
Time Frame: Test of Cure Visit, defined as 14-22 days after the first dose of study drug
Population: The Per Protocol Clinically Evaluable Population included all ITT subjects who took the protocol-defined minimum therapy duration, were dosed with no other antimicrobials (unless allowed by protocol), and had no other major protocol violations
Measure: Number; unit: Participants
Arm/Group | Cethromycin | Clarithromycin
Number analyzed (Participants) | 218 | 208
Participants
  Clinical Cures | 205 | 195
  Clinical Failures | 13 | 13
Statistical Analysis 1: Comparison: Cethromycin vs Clarithromycin; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p > 0.9999, Fisher Exact; Mean Difference (Net) = 0.3, 95% CI [-4.5 to 5.1]

4. Secondary Outcome: Bacteriologic Cures in the Per Protocol Clinically Evaluable Population
Description: as for outcome 2
Time Frame: Test of Cure Visit, defined as 14-22 days after the first dose of study drug.
Population: Includes all Per Protocol Clinically Evaluable subjects that were bacteriologically evaluable (ie., subjects with at least 1 evaluable pathogen) who showed eradication of all evaluable pathogens.
Measure: Number; unit: Participants
Arm/Group | Cethromycin | Clarithromycin
Number analyzed (Participants) | 73 | 69
Participants
  Bacteriologic Cures | 71 | 67

ADVERSE EVENTS:
Time Frame: Reported adverse events were recorded for 30 days after the last dose of study drug for individual subjects.
Description: The safety population was defined as all randomized and dosed subjects with at least one follow up safety assessment.
Arm/Group | Cethromycin | Clarithromycin
Serious Adverse Events (participants affected / at risk) | 13/288 | 9/291
Other Adverse Events (participants affected / at risk) | 55/288 | 37/291
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cethromycin (N=288) | Clarithromycin (N=291)
Acute myocardial infarction (Cardiac disorders) | 4 (4) | 1 (2)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4) | 2 (2)
Empyema (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell lung cancer extensive stage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cethromycin (N=288) | Clarithromycin (N=291)
Diarrhea (Gastrointestinal disorders) | 13 (13) | 12 (13)
Nausea (Gastrointestinal disorders) | 13 (14) | 4 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 7 (8)
Dysgeusia (Nervous system disorders) | 22 (23) | 6 (6)
Headache (Nervous system disorders) | 7 (7) | 8 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other